CLINICAL TRIAL: NCT02009462
Title: Artefill for the Treatment of HIV-associated Facial Lipoatrophy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gerald Pierone, Jr. M.D. (Other)
Collaborators: Suneva Medical, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Gerald Pierone, Jr. M.D., Principle Investigator, AIDS Research and Treatment Center of the Treasure Coast
Organization: AIDS Research and Treatment Center of the Treasure Coast (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARTCTC-01-001
Record Dates: First submitted 2013-12-05; First posted 2013-12-12 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: HIV-facial Lipoatrophy
Keywords: HIV; Facial lipoatrophy
MeSH Terms: interventions — Polymethyl Methacrylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Artefill (Experimental): Four treatment visits using Artefill dermal filler
  Interventions: Drug: Artefill dermal filler

INTERVENTIONS:
Drug: Artefill dermal filler — Four treatment visits will be scheduled at baseline and at weeks 4, 12, and 24. Each treatment session will utilize no more than 8 mL of Artefill and no more than 30 syringes of Artefill.
  Other Names: polymethylmethacrylate (PMMA)

SUMMARY:
Artefill is an injectable facial filler device that is currently approved by the FDA for the correction of nasolabial folds. This study seeks to examine the use of Artefill in the treatment of HIV associated facial lipoatrophy. Facial lipoatrophy (facial fat loss) related to HIV is a stigmatizing condition characterized by loss of facial fat, most notably in the cheeks and temples.

DETAILED DESCRIPTION:
The objectives of this study are:

To evaluate the long-term safety of Artefill injection volumes that are three to four times greater (i.e. up to 30 ml) than the volume indicated in the FDA approved product label (i.e. 8.9 ml)subjects with HIV.

To evaluate any adverse events associated with the use of Artefill. To evaluate the Quality of Life and body image benefit from Artefill treatment in patients with lipoatrophy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female between 18-80 years of age inclusive at the time of signing the informed consent.
2. Subject desires treatment for facial volume loss.
3. Subject has HIV infection with moderated to severe facial lipoatrophy based on the Modified James Scale grades II-IV.
4. Subject has viral load <400 copies/mL.
5. Subject has CD4 lymphocyte counts >200/mm.
6. Subject has documented negative Artefill skin test or has received treatment with Artefill in the past without evidence of hypersensitivity reaction.
7. Subject is willing to withhold additional aesthetic implant therapies (eg, other soft tissue fillers such as Restylane, silicone, Radiesse, Sculptra or implants such as Gortex, Silastic, etc) for the duration of the study.

Exclusion Criteria:

1. Subject has any skin pathology, inflammatory skin disease, or condition that could interfere with the evaluation of the treatment areas.
2. Subject has a history of systemic granulomatous diseases (sarcoid, Wegeners, etc) or connective tissue disease (lupus, dermatomyositis, ect)
3. Subject has history of keloid formation or hypertrophic scarring.
4. Subject has a history of malignancy (other than skin cancer) within 12 months of enrollment. 5.Subject has been treated with systemic corticosteroids(eg, prednisone) or interferon within 1 month prior to study enrollment

6. Subject has thrombocytopenia or a bleeding diathesis. 7. Subject is pregnant, planning to become pregnant, or breastfeeding. 8..Subject has been treated with any of the following within the time intervals specified prior to start of their participation in the study: Bovine collagen-6 months Hyaluronic acid-6 months Calcium hydroxylapatite-6 months Polyacrylamide-at any time Polylactic acid- 6 months Permanent implant grafts at any time. 9. Subject has severe allergies manifested by a history of anaphylaxis or history or presence of multiple severe allergies.

10. Subject has a known hypersensitivity to lidocaine. 11. Subject has a history of allergies to any bovine collagen products. 12. Subject is undergoing or planning to undergo desensitization injections to meat products.

13. Subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.

14. Subject has substance abuse, depression, or other issues that, according to the investigator's judgment, would interfere with conduct of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-12; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Artefill for the Treatment of HIV-Associated Facial Lipoatrophy | 36 months
  To evaluate the effectiveness of Artefill injections as a long-term treatment for human immunodeficiency virus (HIV)-associated facial lipoatrophy over 36 months by assessing changes in the Global Aesthetic Improvement Scale (GAIS) based on pre/post intervention photography.
Artefill for the Treatment of HIV-associated Facial Lipoatrophy | 36 months
  To evaluate the safety of Artefill injections as a long-term treatment for HIV-associated facial lipoatrophy over 36 months by monitoring the incidence of adverse events.

SECONDARY OUTCOMES:
Artefill for the Treatment of HIV-Associated Facial Lipoatrophy | 36 months
  To evaluate the effectiveness of Artefill injections as a long-term treatment for HIV-associated facial lipoatrophy over 36 months by assessing changes in the Modified James Scale grade based on assessment of pre/post intervention photography by 2 blinded physicians.
Artefill for the Treatment of HIV-associated Facial Lipoatrophy | 36 months
  To evaluate the effects of Artefill injections on HIV-associated facial lipoatrophy as evidenced by the subject satisfaction questionnaire.
Artefill for the Treatment of HIV-associated Facial Lipoatrophy | 36 months
  To evaluate the effects of Artefill injections on the subject's psychological well-being using the Medical Outcomes study-HIV (MOS-HIV)assessment.
Artefill for the Treatment of HIV-associated Facial Lipoatrophy | 36 months
  To evaluate the acceptability and tolerability of Artefill injections as reported by subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Pierone, Jr., M.D, Principal Investigator — AIDS Research and Treatment Center of the Treasure Coast
Locations (1):
- Whole Family Health Center, Vero Beach, Florida, United States